CLINICAL TRIAL: NCT01436656
Title: A Phase I, Multicenter, Open-label, Dose-escalation Study of Oral LGX818 in Adult Patients With Locally Advanced or Metastatic BRAF Mutant Melanoma
Brief Title: A Phase I Study of Oral LGX818 in Adult Patients With Advanced or Metastatic BRAF Mutant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGX818X2101; C4221010 (Other: Alias Study Number); 2011-000556-42 (EudraCT Number)
Record Dates: First submitted 2011-04-14; First posted 2011-09-20 (Estimated); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Melanoma and Metastatic Colorectal Cancer
Keywords: BRAF mutant,; BRAF mutated,; melanoma,; metastatic,; advanced,; RAF kinase inhibitor; BRAF V600 mutation
MeSH Terms: conditions — Melanoma; Colorectal Neoplasms; Neoplasm Metastasis | interventions — encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- LGX818 - Dose escalation (Experimental)
  Interventions: Drug: LGX818
- LGX818 - Dose Expansion at MTD or RP2D (Experimental)
  Interventions: Drug: LGX818

INTERVENTIONS:
Drug: LGX818

SUMMARY:
CLGX818X2101 is a first-time in-human, phase I study to establish the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of daily administered LGX818 (daily, twice daily and/or every-other-day), a RAF kinase inhibitor. Patients with locally advanced or metastatic melanoma harboring the BRAF V600 mutation (during dose escalation phase and expansion phase) and patients with metastatic colorectal cancer harboring the BRAF V600 mutation (during the expansion phase) will be enrolled. The study consists of a dose escalation part were cohorts of patients will receive escalating oral doses of LGX818, followed by a safety dose expansion part were patients will be treated with oral dose of LGX818 given at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

For the dose escalation phase:

1. Histologically confirmed diagnosis of locally advanced or metastatic melanoma (stage IIIB to IV per American Joint Committee on Cancer [AJCC]). For the dose expansion phase: (i) Histologically confirmed diagnosis of locally advanced or metastatic melanoma (stage IIIB to IV per American Joint Committee on Cancer [AJCC]), or (ii) confirmed diagnosis and non-resectable advanced metastatic colorectal cancer (mCRC) for which no further effective standard therapy exists.
2. Written documentation of BRAF V600E mutation, or any other BRAF V600 mutation.
3. Evidence of measurable disease

Exclusion Criteria:

1. Previous therapy with a MEK inhibitor.
2. Symptomatic or untreated leptomeningeal disease.
3. Symptomatic or untreated brain metastasis.Patients previously treated for these conditions that are asymptomatic in the absence of corticosteroid therapy are allowed to enroll. Brain metastasis must be stable with verification by imaging.
4. Known acute or chronic pancreatitis.
5. Clinically significant cardiac disease
6. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LGX818
7. Previous or concurrent malignancy. Exceptions to this exclusion criteria include: adequately treated basal cell or squamous cell skin cancer; in situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 3 years prior to study entry; or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry.
8. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
9. History of thromboembolic or cerebrovascular events within the last 6 months

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2012-10-01 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (5):
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Australia (3):
  - Western Sydney Local Health District, Westmead, New South Wales
  - Westmead Hospital- Redbank Rd, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
- France (5):
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse, Haute-garonne
  - Institut Gustave Roussy, Villejuif, ILE de France - VAL de Marne (94)
  - Institut Gustave Roussy, Villejuif, VAL DE Marne
  - Institut Gustave Roussy, Villejuif, Val-de-marne
  - Institut Gustave Roussy, Villejuif
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan
- Oslo Myeloma Center - PPDS, Oslo, Norway
- Spain (6):
  - Hospital Clinic de Barcelona, Badalona
  - Hospital General Vall d'Hebron, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario HM Sanchinarro_CIOCC, Madrid
  - START MADRID_Hospital Universitario HM Sanchinarro - CIOCC, Madrid
- Switzerland (2):
  - Kantonsspital Graubünden, Chur, Graubünden (DE)
  - Universität Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 107 participants (54 in dose escalation and 53 in dose expansion) were enrolled in this study.
Groups:
- 50 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 50 milligram (mg) encorafenib (LGX818) orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 100 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 100 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 150 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 150 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 75 mg Encorafenib BID: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 75 mg encorafenib orally twice daily (BID) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 300 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 300 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 150 mg Encorafenib BID: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 150 mg encorafenib twice daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 200 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 200 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 100 mg Encorafenib BID: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 100 mg encorafenib twice daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 450 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 450 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 550 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 550 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 700 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 700 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Mel Naive 300 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations naive to a selective BRAF inhibitor received 300 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Mel Naive 450 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations naive to a selective BRAF inhibitor received 450 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Mel Pre-treated: 300 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations pre-treated to a selective BRAF inhibitor received 300 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Mel Pre-treated: 450 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations pre-treated to a selective BRAF inhibitor received 450 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Mel Stepwise: 450 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations received 450 mg encorafenib orally QD in a two-step manner in each 28-day treatment cycle until disease progression, withdrawal of consent or unacceptable toxicity.
- Metastatic Colorectal Cancer: 300 mg Encorafenib: Participants with metastatic colorectal cancer received 300 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or unacceptable toxicity.
- Metastatic Colorectal Cancer: 450 mg Encorafenib: Participants with metastatic colorectal cancer received 450 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or unacceptable toxicity.
Period: Dose Escalation
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Started | 4 | 10 | 6 | 3 | 5 | 4 | 4 | 5 | 6 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 6 | 5 | 3 | 1 | 2 | 3 | 2 | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 1 | 0 | 4 | 2 | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative problems | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — New anti-cancer therapy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 (Participants enrolled in dose expansion phase.) | 6 (Participants enrolled in dose expansion phase.) | 2 (Participants enrolled in dose expansion phase.) | 16 (Participants enrolled in dose expansion phase.) | 2 (Participants enrolled in dose expansion phase.) | 6 (Participants enrolled in dose expansion phase.) | 12 (Participants enrolled in dose expansion phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 8 | 2 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 1 | 8 | 0 | 4 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — New cancer therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants from the full analysis set (all participants who received at least one dose of encorafenib) who had at least one valid post-baseline safety assessment.
Groups:
- 50 mg of Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 50 mg encorafenib (LGX818) orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity
- Total: Total of all reporting groups
Arm/Group | 50 mg of Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib | Total
Number analyzed (Participants) | 4 | 10 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2 | 9 | 6 | 2 | 16 | 2 | 6 | 12 | 107
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 44 years | 1 | 3 | 1 | 1 | 4 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 7 | 1 | 0 | 1 | 27
  Between 45 and 64 years | 3 | 4 | 3 | 1 | 0 | 5 | 1 | 1 | 2 | 4 | 1 | 7 | 3 | 0 | 4 | 1 | 4 | 7 | 51
  >=65 years | 0 | 3 | 2 | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 5 | 0 | 2 | 4 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 0 | 2 | 0 | 1 | 2 | 4 | 1 | 1 | 4 | 1 | 1 | 13 | 1 | 3 | 7 | 48
  Male | 2 | 7 | 4 | 3 | 2 | 5 | 4 | 2 | 2 | 4 | 1 | 5 | 5 | 1 | 3 | 1 | 3 | 5 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 10 | 6 | 3 | 4 | 4 | 5 | 4 | 6 | 4 | 2 | 6 | 5 | 1 | 16 | 2 | 6 | 12 | 100
  Others | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) During Dose Escalation Phase
Description: DLT= Adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within first 28 days of treatment with encorafenib and met any of following criteria: >=grade (G)3 neutropenia or thrombocytopenia for >7 days; G4 thrombocytopenia; febrile neutropenia; >=G3 serum creatinine, blood bilirubin; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) and lipase and/or serum amylase (>=G3 for > 7 consecutive days or G4); >=G3 ALT or AST and >=G2 blood bilirubin; >=G3 persistent hypertension with more than one drug or more intensive therapy or cardiac disorders or AE excluding on-target side-effect that is manageable; G3 fatigue/asthenia for >7 consecutive days; >= G3 vomiting or nausea or diarrhea lasting more than 48 hours despite treatment; >=G3 pancreatitis, rash/photosensitivity (G3 for > 7 consecutive days despite skin toxicity treatment or G4); G3 or G4 eye disorders.
Time Frame: Up to 28 days
Population: Dose-Determining Set (DDS) consisted of all participants from the safety set who either met the following minimum exposure (received at least 75% of the planned doses of encorafenib in Cycle 1; observed for at least 1 cycle and considered to have sufficient safety data to conclude that a DLT did not occur in cycle 1) and had completed scheduled safety evaluations or experienced a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- 50 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 50 milligram (mg) encorafenib orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 4 | 9 | 6 | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 2
Participants | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2

2. Primary Outcome: Number of Participants With DLT During Dose Expansion Phase
Description: as for outcome 1
Time Frame: Up to 28 days
Population: DDS consisted of all participants from the safety set who either met the following minimum exposure criterion (received at least 75% of the planned doses of encorafenib in Cycle 1; observed for at least 1 cycle and considered to have sufficient safety data to conclude that a DLT did not occur in cycle 1) and had completed scheduled safety evaluations or experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 9 | 2 | 1 | 13 | 2 | 5 | 12
Participants | 2 | 2 | 0 | 4 | 1 | 0 | 3

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) During Dose Escalation Phase
Description: An AE was defined as the appearance of (or worsening of any pre-existing) undesirable signs, symptoms, or medical conditions. An SAE was defined as one of the following: fatal or life-threatening; resulted in significant disability/incapacity; congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization unless for routine treatment, elective or pre-planned treatment for a pre-existing condition, treatment on an emergency outpatient basis, social reasons and respite care in the absence of any deterioration in the participants general condition, any SAEs that were expected due to the condition being treated.
Time Frame: From start of study treatment until 30 days after last dose of study treatment (maximum of 556.1 weeks of treatment exposure)
Population: Safety set included all participants who received at least one dose of encorafenib and had at least one valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 4 | 10 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Participants
  Adverse Events (AEs) | 4 | 10 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
  Serious Adverse Events (SAEs) | 3 | 7 | 3 | 2 | 4 | 2 | 4 | 2 | 2 | 3 | 1

4. Secondary Outcome: Number of Participants With AEs and SAEs During Dose Expansion Phase
Description: as for outcome 3
Time Frame: From start of study treatment until 30 days after last dose of study treatment (maximum of 257.3 weeks and 114.6 weeks of treatment exposure for melanoma participants and mCRC participants respectively)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 9 | 6 | 2 | 16 | 2 | 6 | 12
Participants
  Adverse Events (AEs) | 9 | 6 | 2 | 16 | 2 | 6 | 12
  Serious Adverse Events (SAEs) | 2 | 4 | 2 | 9 | 2 | 3 | 6

5. Secondary Outcome: Progression Free Survival (PFS): Dose Escalation Phase
Description: PFS was defined as time from date of first study treatment intake to date of first documented disease progression (PD) or death due to any cause. If a participant did not have an event, data censoring was done at the date of last adequate tumor assessment. PD was defined for target disease as at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study (this included baseline sum if that was smallest on study), sum also demonstrated absolute increase of greater than or equal to (>=) 5 mm, or appearance of >=1 new lesions. For non-target disease: PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion was also considered PD. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until first documentation of PD or death due to any cause or censoring date (maximum of 556.1 weeks of treatment exposure)
Population: Full Analysis Set (FAS) included all participants who received at least one dose of encorafenib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 4 | 10 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Months | 75.0 [19.4 to 99.4] | 10.0 [0.3 to 44.5] | 50.0 [11.8 to 88.2] | 33.3 [0.8 to 90.6] | 50.0 [6.8 to 93.2] | 40.0 [5.3 to 85.3] | 0.0 [0.0 to 52.2] | 75.0 [19.4 to 99.4] | 33.3 [4.3 to 77.7] | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 84.2]

6. Secondary Outcome: PFS: Dose Expansion Phase
Description: PFS was defined as time from date of first study treatment intake to date of first documented PD or death due to any cause. If a participant did not have an event, data censoring was done at the date of last adequate tumor assessment. PD was defined for target disease as at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study (this included baseline sum if that was smallest on study), sum also demonstrated absolute increase of >= 5 mm, or appearance of >=1 new lesions. For non-target disease: PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion was also considered PD. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until first documentation of PD or death due to any cause or censoring date (maximum of 257.3 weeks and 114.6 weeks of treatment exposure for melanoma participants and mCRC participants respectively)
Population: FAS included all participants who received at least one dose of encorafenib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 9 | 6 | 2 | 16 | 2 | 6 | 12
Months | 16.5 [7.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 19.3 [7.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 0.6 [0.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 2.0 [1.6 to 3.7] | 20.1 [10.9 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 4.5 [2.3 to 7.2] | 4.0 [1.8 to 5.5]

7. Secondary Outcome: Duration of Response (DOR): Dose Escalation Phase
Description: DOR was defined as the time from first observation of response CR or partial response [PR]) to the first time of progression or death. CR was defined as complete disappearance of all target and non-target lesions, and sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. For target disease, PD=at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study, sum also demonstrated absolute increase of >= 5 mm, or appearance of >=1 new lesions. For non-target disease: PD=unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion.
Time Frame: From first observation of response until first time of PD or death due to any cause (Maximum of 556.1 weeks of treatment exposure)
Population: FAS included all participants who received at least one dose of encorafenib. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Only participants with complete or partial response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 3 | 1 | 3 | 1 | 2 | 2 | 0 | 3 | 2 | 1 | 0
Months | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. |  | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. |

8. Secondary Outcome: Time to Response (TTR): Dose Escalation Phase
Description: TTR was defined as the time from date of treatment until first documented response (CR or PR). CR was defined as complete disappearance of all target and non-target lesions sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants who did not achieve a confirmed PR or CR, were censored at last adequate tumor assessment date when they did not progress (including deaths not due to underlying disease) or at maximum follow-up (from study start to study end date) when participant had an event for progression-free survival. Individual participant data have been reported for this outcome measure.
Time Frame: From date of start of treatment until CR or PR or censoring date (maximum of 556.1 weeks of treatment exposure)
Population: FAS included all participants who received at least one dose of encorafenib.'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Only participants with complete or partial response were included in the analysis.
Measure: Number; unit: Days
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 3 | 1 | 3 | 1 | 2 | 2 | 0 | 3 | 2 | 1 | 0
Days
  Participant 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 1 | 57 |  |  |  |  |  |  |  |  |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 2 | 952 |  |  |  |  |  |  |  |  |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 3 | 22 |  |  |  |  |  |  |  |  |  |
  Participant 4: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 4 |  | 55 |  |  |  |  |  |  |  |  |
  Participant 5: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 5 |  |  | 897 |  |  |  |  |  |  |  |
  Participant 6: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 6 |  |  | 21 |  |  |  |  |  |  |  |
  Participant 7: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 7 |  |  | 72 |  |  |  |  |  |  |  |
  Participant 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 8 |  |  |  |  | 27 |  |  |  |  |  |
  Participant 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 9 |  |  |  |  | 57 |  |  |  |  |  |
  Participant 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participant 10 |  |  |  |  |  |  |  |  | 57 |  |
  Participant 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participant 11 |  |  |  |  |  |  |  |  | 627 |  |
  Participant 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Participant 12 |  |  |  |  |  |  |  |  |  | 56 |
  Participant 13: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 13 |  |  |  | 28 |  |  |  |  |  |  |
  Participant 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Participant 14 |  |  |  |  |  | 280 |  |  |  |  |
  Participant 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Participant 15 |  |  |  |  |  | 22 |  |  |  |  |
  Participant 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 16 |  |  |  |  |  |  |  | 22 |  |  |
  Participant 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 17 |  |  |  |  |  |  |  | 29 |  |  |
  Participant 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 18 |  |  |  |  |  |  |  | 727 |  |  |

9. Secondary Outcome: DOR: Dose Expansion Phase
Description: DOR was defined as the time from first observation of response (CR or PR] to the first time of progression or death. CR was defined as complete disappearance of all target and non-target lesions and sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to (<10 mm. PR defined as at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. For target disease, PD=at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study, sum also demonstrated absolute increase of >= 5 mm, or appearance of >=1 new lesions. For non-target disease: PD=unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion.
Time Frame: From first observation of response until first time of PD or death due to any cause (maximum of 257.3 weeks and 114.6 weeks of treatment exposure for melanoma participants and mCRC participants respectively)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 7 | 2 | 0 | 4 | 1 | 1 | 0
Months | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. |  | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. |

10. Secondary Outcome: TTR: Dose Expansion Phase
Description: as for outcome 8
Time Frame: From date of start of treatment until CR or PR or censoring date (maximum of 257.3 weeks and 114.6 weeks of treatment exposure for melanoma participants and mCRC participants respectively)
Population: FAS included all participants who received at least one dose of encorafenib. 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Only participants with complete or partial response were included in the analysis.
Measure: Number; unit: Days
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 7 | 2 | 0 | 4 | 1 | 1 | 0
Days
  Participant 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 1 | 211 |  |  |  |  |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 2 | 22 |  |  |  |  |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 3 | 23 |  |  |  |  |  |
  Participant 4: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 4 | 22 |  |  |  |  |  |
  Participant 5: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 5 | 56 |  |  |  |  |  |
  Participant 6: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 6 | 23 |  |  |  |  |  |
  Participant 7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant 7 | 56 |  |  |  |  |  |
  Participant 8: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Participant 8 |  | 78 |  |  |  |  |
  Participant 9: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Participant 9 |  | 111 |  |  |  |  |
  Participant 10: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 10 |  |  |  | 391 |  |  |
  Participant 11: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 11 |  |  |  | 22 |  |  |
  Participant 12: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 12 |  |  |  | 32 |  |  |
  Participant 13: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participant 13 |  |  |  | 28 |  |  |
  Participant 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participant 14 |  |  |  |  | 25 |  |
  Participant 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Participant 15 |  |  |  |  |  | 53 |

11. Secondary Outcome: Overall Survival (OS): Dose Expansion Phase
Description: Overall survival was defined as the time from the date of first study treatment to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until date of death or censoring date (maximum of 257.3 weeks and 114.6 weeks of treatment exposure for melanoma participants and mCRC participants respectively)
Population: FAS included all participants who received at least one dose of encorafenib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 9 | 6 | 2 | 16 | 2 | 6 | 12
Months | NA [11.6 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 12.5 [7.7 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events | NA [2.4 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 9.5 [3.7 to 13.2] | NA [30.7 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 7.2 [5.6 to 10.5] | 8.0 [4.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events

12. Secondary Outcome: Maximum Observed Plasma Concentration of LGX818: Dose Escalation Phase
Time Frame: Pre-dose (0 hour), 0.5, 3, 4, 6, 8, 10 (only for BID arms), 24 hours post dose on Day 1 and 15 of Cycle 1 (each cycle=28 days)
Population: Pharmacokinetic Analysis Set (PAS) consisted of all participants who had at least one blood sample providing evaluable pharmacokinetic (PK) data. Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- 50 mg Encorafenib QD (Capsules): Participants received 50 mg of LGX818 capsule orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 50 mg Encorafenib QD (Microemulsion): Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 50 mg encorafenib (LGX818) as microemulsion orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 100 mg Encorafenib QD (Capsules): Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 100 mg encorafenib (LGX818) capsules orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 100 mg Encorafenib QD (Microemulsion): Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 100 mg encorafenib (LGX818) as microemulsion orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- 100 mg of Encorafenib BID (Microemulsion): Participants received 200 mg of LGX818 orally once daily for each 28-day treatment cycle until disease progression, withdrawal of consent, unacceptable toxicity, or termination of treatment, followed by a 30-day safety assessment for toxicity.
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg of Encorafenib BID (Microemulsion) | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Nanogram per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 2 | 4 | 5 | 5 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 970 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed | 846 (82.92) | 1630 (42.36) | 1020 (49.06) | 1570 (28.82) | 733 (46.32) | 1850 (28.06) | 1200 (28.06) | 3310 (42.54) | 2510 (58.15) | 5970 (56.35) | 5360 (36.87) | 8980 (13.5)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 4 | 5 | 5 | 3 | 4 | 5 | 4 | 4 | 6 | 3 | 2
  Cycle 1 Day 15 | 465 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed | 334 (57.7) | 959 (25.19) | 949 (27.4) | 1300 (29.08) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 1300 (1220) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 2920 (34.41) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 3950 (49.12) | 4170 (48.94) | NA (NA) — Data could not be estimated as values were below limit of quantitation.

13. Secondary Outcome: Time Point of Maximum Concentration (Tmax) of LGX818: Dose Escalation Phase
Time Frame: as for outcome 12
Population: PAS consisted of all participants who had at least one blood sample providing evaluable pharmacokinetic (PK) data. Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Median (Full Range); unit: Hours
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 2 [2 to 2] | 0.5 [0.167 to 0.500] | 2 [0.5 to 2] | 2 [0.5 to 2] | 2 [0.517 to 3.95] | 2.02 [2 to 4.08] | 2 [2 to 2] | 2 [2 to 2.08] | 2 [2 to 8] | 1.25 [0.5 to 2.25] | 2 [2 to 2.33] | 2 [2 to 2.07] | 2.04 [2 to 2.08]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 4 | 5 | 5 | 3 | 4 | 5 | 4 | 4 | 6 | 3 | 2
  Cycle 1 Day 15 | 2 [2 to 2] | 0.5 [0.5 to 2] | 2.99 [2 to 4] | 0.5 [0.5 to 0.533] | 2 [0.5 to 2.03] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 2 [2 to 2.17] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 2 [2 to 2.02] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 2 [0.5 to 2] | 2 [2 to 2] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation.

14. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinf) of LGX818: Dose Escalation Phase
Description: AUC (inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*Nanogram per milliliter
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Hours*Nanogram per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 3 | 4 | 3 | 4 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 5470 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 2340 (70.37) | 7660 (83.44) | 5050 (39.57) | 9520 (20.11) | 2220 (53.66) | 9910 (26.24) | 4410 (69.51) | 20000 (33.36) | 8940 (50) | 33100 (70.34) | 31900 (45.51) | 64400 (1.75)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 4 | 3 | 6 | 3 | 4 | 5 | 4 | 4 | 6 | 3 | 2
  Cycle 1 Day 15 | 2700 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 1130 (20.1) | 5380 (36.87) | 2900 (37.88) | 4830 (11.11) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 5080 (35.87) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 10200 (53.84) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 13200 (34.77) | 15600 (36.58) | NA (NA) — Data could not be estimated as values were below limit of quantitation.

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Tau (AUCtau) of LGX818: Dose Escalation Phase
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*Nanogram per milliliter
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Hours*Nanogram per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 5360 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 2330 (69.89) | 7610 (82.98) | 5010 (39.39) | 9400 (20.06) | 3210 (92.21) | 9860 (26.5) | 4780 (52.49) | 20300 (29.06) | 8690 (49.73) | 32800 (69.05) | 31700 (45.33) | 63900 (1.41)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 4 | 3 | 6 | 3 | 4 | 5 | 4 | 4 | 6 | 3 | 2
  Cycle 1 Day 15 | 2660 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 1120 (19.67) | 5330 (36.58) | 2890 (37.55) | 4750 (12.25) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 5060 (35.79) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 10100 (53.35) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 13100 (34.85) | 15300 (36.38) | NA (NA) — Data could not be estimated as values were below limit of quantitation.

16. Secondary Outcome: Elimination Half-life (t1/2) of LGX818: Dose Escalation Phase
Description: t1/2 was the time measured for the plasma concentration to decrease by one half. Terminal phase half-life expressed in hours (hr).
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 3 | 4 | 3 | 4 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 4.38 [4.38 to 4.38] | 3.77 [3.57 to 4.44] | 3.47 [3.38 to 3.88] | 3.7 [3.32 to 3.96] | 3.66 [3.09 to 4.5] | 2.82 [2.02 to 3.84] | 3.3 [2.56 to 3.58] | 2.53 [1.69 to 2.68] | 3.42 [2.84 to 4.77] | 2.16 [2.16 to 2.42] | 2.92 [2.32 to 4.98] | 3.32 [3.28 to 3.61] | 3.25 [2.96 to 3.53]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 4 | 3 | 6 | 3 | 4 | 5 | 4 | 4 | 6 | 3 | 2
  Cycle 1 Day 15 | 4.14 [4.14 to 4.14] | 3.71 [3.66 to 5.63] | 3.99 [3.22 to 4.05] | 3.61 [3.26 to 4.1] | 3.65 [3.43 to 7.47] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 3.13 [2.95 to 3.22] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 3.57 [1.61 to 4.06] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 3.19 [2.82 to 3.56] | 3.25 [2.96 to 8] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation.

17. Secondary Outcome: Apparent Total Plasma Clearance of Drug (CL/F) of LGX818: Dose Escalation Phase
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Liter/hour
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 9.14 (NA) — The geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 21.3 (70.37) | 13 (83.44) | 19.8 (39.57) | 15.8 (20.11) | 33.8 (53.66) | 20.2 (26.24) | 22.7 (69.51) | 15 (33.36) | 16.8 (50) | 13.6 (70.34) | 17.2 (45.51) | 10.9 (1.75)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 3 | 5 | 6 | 2 | 4 | 5 | 4 | 4 | 6 | 3 | 2
  Cycle 1 Day 15 | 18.8 (NA) — The geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 44.7 (19.67) | 18.8 (36.58) | 34.6 (37.55) | 31.5 (12.25) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 39.5 (35.79) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 29.6 (53.35) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 34.3 (34.85) | 36 (36.38) | NA (NA) — Data could not be estimated as values were below limit of quantitation.

18. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of LGX818: Dose Escalation Phase
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | 50 mg Encorafenib QD (Capsules) | 50 mg Encorafenib QD (Microemulsion) | 100 mg Encorafenib QD (Capsules) | 100 mg Encorafenib QD (Microemulsion) | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 1 | 3 | 5 | 5 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Liter
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 5 | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 6 | 5 | 2
  Cycle 1 Day 1 | 57.8 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 120 (56.42) | 67 (79.38) | 104 (35.34) | 84.5 (28.15) | 116 (27.23) | 91.9 (39.62) | 73.8 (39.95) | 76.5 (33.65) | 53.9 (49.07) | 60.5 (53.31) | 84.8 (41.99) | 50.7 (10.87)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5 | 4 | 6 | 5 | 2
  Cycle 1 Day 15 | 112 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 274 (7.68) | 103 (36.42) | 182 (33.22) | 188 (43.23) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 177 (31) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 128 (12.49) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 157 (38.55) | 221 (75.92) | NA (NA) — Data could not be estimated as values were below limit of quantitation.

19. Secondary Outcome: Number of Participants According to Tumor Response Per RECIST Criteria- Dose Escalation
Description: Tumor response included: CR, PR, stable disease and disease progression (PD). CR=complete disappearance of all target and non-target lesions sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm. PR=at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease=neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. For target disease, PD=at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study, sum also demonstrated absolute increase of >= 5 mm, or appearance of >=1 new lesions. For non-target disease: PD=unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion.
Time Frame: as for outcome 5
Population: FAS included all participants who received at least one dose of encorafenib.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Encorafenib QD | 100 mg Encorafenib QD | 150 mg Encorafenib QD | 75 mg Encorafenib BID | 200 mg Encorafenib QD | 100 mg Encorafenib BID | 300 mg Encorafenib QD | 150 mg Encorafenib BID | 450 mg Encorafenib QD | 550 mg Encorafenib QD | 700 mg Encorafenib QD
Number analyzed (Participants) | 4 | 10 | 6 | 3 | 4 | 5 | 5 | 4 | 6 | 5 | 2
Participants
  Complete Response (CR) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Partial Response (PR) | 2 | 1 | 3 | 1 | 1 | 2 | 0 | 2 | 2 | 1 | 0
  Stable Disease (SD) | 0 | 5 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 1
  Progressive Disease (PD) | 1 | 2 | 2 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 0

20. Secondary Outcome: Maximum Observed Plasma Concentration of LGX818: Dose Expansion Phase
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 1 | 10
Nanogram per milliliter
  Cycle 1 Day 1 | 4310 (31.6) | 5650 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 7790 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 6580 (34.24) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 1340 | 8380 (32.93)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 1060 (41.1) |  |  | 5590 (22.56) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 5650 (79.98)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 0 | 0 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 2050 (43.71) |  |  | 4960 (32.64) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 1040 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 5130 (48.81)

21. Secondary Outcome: Vz/F of LGX818: Dose Expansion Phase
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: PAS consisted of all participants who had at least one blood sample providing evaluable pharmacokinetic (PK) data. 'Overall Number of Participants Analyzed' signifies number of participants with evaluable data for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 0 | 1 | 10 | 2 | 1 | 10
Liter
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 0 | 1 | 10 | 2 | 0 | 10
  Cycle 1 Day 1 | 79.1 (29.82) |  | 25.3 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 59.7 (35.42) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 44.6 (26.6)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 219 (41.9) |  |  | 66.1 (23.07) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 70 (40.28)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 0 | 0 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 243 (79) |  |  | 130 (20.81) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 194 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 110 (32.51)

22. Secondary Outcome: Tmax of LGX818: Dose Expansion Phase
Description: Tmax was the time required to reach the maximum plasma concentration (Cmax). First observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in hours (hr).
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 1 | 10
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 0 | 10
  Cycle 1 Day 1 | 1.97 [1.95 to 1.97] | 2.08 [2.08 to 2.08] | 3.97 [3.97 to 3.97] | 2 [0.5 to 2.12] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. |  | 2 [0.667 to 4]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 1.92 [1.9 to 1.98] |  |  | 1.93 [0.5 to 2.07] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. |  | 2 [0.5 to 2]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 1 | 1 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 1.9 [1.88 to 1.97] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 2 [0.5 to 2.3] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 4 [4 to 4] | 2 [1.97 to 2.08]

23. Secondary Outcome: AUCinf of LGX818: Dose Expansion Phase
Description: as for outcome 14
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*Nanogram per milliliter
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 0 | 1 | 10 | 2 | 1 | 10
Hours*Nanogram per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 0 | 1 | 10 | 2 | 0 | 10
  Cycle 1 Day 1 | 18200 (32.37) |  | 70900 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 33300 (39.98) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 54400 (42.97)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 4290 (30.9) |  |  | 16600 (23.69) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 16400 (34.68)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 0 | 0 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 2050 (43.71) |  |  | 4960 (32.64) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 1040 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 17300 (38.06)

24. Secondary Outcome: AUCtau of LGX818: Dose Expansion Phase
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 1 | 10
hours*nanogram per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 0 | 10
  Cycle 1 Day 1 | 18100 (32.22) | 35300 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 69300 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 33200 (39.86) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 54400 (42.97)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 4290 (30.9) |  |  | 16600 (23.69) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 16400 (34.67)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 0 | 0 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 7380 (60.51) |  |  | 17600 (25.65) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 10400 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 17300 (37.9)

25. Secondary Outcome: t1/2 of LGX818: Dose Expansion Phase
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 1 | 10
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 1 | 1 | 10 | 2 | 0 | 10
  Cycle 1 Day 1 | 3.36 [3 to 3.65] | 4.04 [4.04 to 4.04] | 4.14 [4.14 to 4.14] | 3.07 [2.61 to 3.38] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. |  | 3.63 [2.59 to 6.44]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 2.41 [1.69 to 2.47] |  |  | 1.66 [1.61 to 1.81] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. |  | 1.76 [1.62 to 1.98]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 0 | 0 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 4.33 [3.47 to 4.75] |  |  | 3.37 [2.87 to 4.24] | NA [NA to NA] — Data could not be estimated as values were below limit of quantitation. | 4.51 [4.51 to 4.51] | 3.13 [1.73 to 4.42]

26. Secondary Outcome: CL/F of LGX818: Dose Expansion Phase
Time Frame: Predose (0 hour), 0.5, 2, 4, 6, 8, 24 hours post dose on Day 1,8 and 15 of Cycle 1 (cycle=28 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 3 | 0 | 1 | 10 | 2 | 1 | 10
liter/hour
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 0 | 1 | 10 | 2 | 0 | 10
  Cycle 1 Day 1 | 16.5 (32.37) |  | 4.23 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 13.5 (39.98) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 8.27 (42.97)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 0 | 0 | 5 | 2 | 0 | 5
  Cycle 1 Day 8 | 70.1 (30.98) |  |  | 27.2 (23.63) | NA (NA) — Data could not be estimated as values were below limit of quantitation. |  | 27.4 (34.67)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 0 | 0 | 7 | 2 | 1 | 7
  Cycle 1 Day 15 | 40.7 (60.51) |  |  | 25.6 (25.65) | NA (NA) — Data could not be estimated as values were below limit of quantitation. | 29.9 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 26 (37.9)

27. Secondary Outcome: Number of Participants According to BRAF V600 Mutation Status at Baseline: Dose Expansion
Description: Number of participants according to BRAF V600 mutation status as V600E (i.e., mutation of the BRAF gene in which valine [V] was substituted by glutamic acid [E] at amino acid 600) or other is reported in this outcome measure.
Time Frame: (Baseline) last non-missing value prior to the first dose (Baseline)
Population: FAS included all participants who received at least one dose of Encorafenib
Measure: Count of Participants; unit: Participants
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 9 | 6 | 2 | 16 | 2 | 6 | 12
Participants
  V600E | 8 | 5 | 1 | 16 | 1 | 6 | 12
  Others | 1 | 1 | 1 | 0 | 1 | 0 | 0

28. Secondary Outcome: Number of Participants According to Tumor Response Per RECIST Criteria: Dose Expansion
Description: umor response included: CR, PR, stable disease and disease progression (PD). CR=complete disappearance of all target and non-target lesions sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm. PR=at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease=neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. For target disease, PD=at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study, sum also demonstrated absolute increase of >= 5 mm, or appearance of >=1 new lesions. For non-target disease: PD=unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion.
Time Frame: as for outcome 6
Population: FAS included all participants who received at least one dose of encorafenib.
Measure: Count of Participants; unit: Participants
Arm/Group | Mel Naive 300 mg Encorafenib | Mel Naive 450 mg Encorafenib | Mel Pre-treated: 300 mg Encorafenib | Mel Pre-treated: 450 mg Encorafenib | Mel Stepwise: 450 mg Encorafenib | Metastatic Colorectal Cancer: 300 mg Encorafenib | Metastatic Colorectal Cancer: 450 mg Encorafenib
Number analyzed (Participants) | 9 | 6 | 2 | 16 | 2 | 6 | 12
Participants
  Complete Response (CR) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 6 | 2 | 0 | 4 | 1 | 1 | 0
  Stable Disease (SD) | 0 | 1 | 0 | 2 | 1 | 3 | 8
  Progressive Disease (PD) | 1 | 0 | 2 | 8 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: From start of study treatment until 30 days after last dose of study treatment (maximum of 556.1 weeks of treatment exposure) for Dose escalation arms and (maximum of 257.3 weeks and 114.6 weeks of treatment exposure for melanoma participants and mCRC participants respectively) for Dose expansion arms.
Description: Same event may appear as both non-SAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and non-serious in another participants, or one participant may have experienced both serious and non-serious event during the study.
Groups:
- Dose Escalation: 50 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 50 mg encorafenib (LGX818) orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity
- Dose Escalation: 100 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 100 mg encorafenib orally once daily (QD) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity
- Dose Escalation:150 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 150 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 75 mg Encorafenib BID: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 75 mg encorafenib orally twice daily (BID) in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 200 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 200 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 100 mg Encorafenib BID: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 100 mg encorafenib twice daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 300 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 300 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 150 mg Encorafenib BID: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 150 mg encorafenib twice daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 450 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 450 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 550 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 550 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Escalation: 700 mg Encorafenib QD: Participants with advanced or metastatic melanoma harboring BRAF V600 (E, K, D, R) mutations received 700 mg encorafenib orally once daily in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Expansion: Mel Naive 300 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations naive to a selective BRAF inhibitor received 300 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Expansion: Mel Naive 450 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations naive to a selective BRAF inhibitor received 450 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Expansion: Mel Pre-treated 300 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations pre-treated to a selective BRAF inhibitor received 300 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Expansion: Mel Pre-treated 450 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations pre-treated to a selective BRAF inhibitor received 450 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or, unacceptable toxicity.
- Dose Expansion: Mel Stepwise 450 mg Encorafenib: Participants with advanced melanoma harboring BRAF V600 (E, K, D, R) mutations received 450 mg encorafenib orally QD in a two-step manner in each 28-day treatment cycle until disease progression, withdrawal of consent or unacceptable toxicity.
- Dose Expansion: Metastatic Colorectal Cancer 300 mg Encorafenib: Participants with metastatic colorectal cancer received 300 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or unacceptable toxicity.
- Dose Expansion: Metastatic Colorectal Cancer 450 mg Encorafenib: Participants with metastatic colorectal cancer received 450 mg encorafenib orally QD in each 28-day treatment cycle until disease progression, withdrawal of consent or unacceptable toxicity.
Arm/Group | Dose Escalation: 50 mg Encorafenib QD | Dose Escalation: 100 mg Encorafenib QD | Dose Escalation:150 mg Encorafenib QD | Dose Escalation: 75 mg Encorafenib BID | Dose Escalation: 200 mg Encorafenib QD | Dose Escalation: 100 mg Encorafenib BID | Dose Escalation: 300 mg Encorafenib QD | Dose Escalation: 150 mg Encorafenib BID | Dose Escalation: 450 mg Encorafenib QD | Dose Escalation: 550 mg Encorafenib QD | Dose Escalation: 700 mg Encorafenib QD | Dose Expansion: Mel Naive 300 mg Encorafenib | Dose Expansion: Mel Naive 450 mg Encorafenib | Dose Expansion: Mel Pre-treated 300 mg Encorafenib | Dose Expansion: Mel Pre-treated 450 mg Encorafenib | Dose Expansion: Mel Stepwise 450 mg Encorafenib | Dose Expansion: Metastatic Colorectal Cancer 300 mg Encorafenib | Dose Expansion: Metastatic Colorectal Cancer 450 mg Encorafenib
All-Cause Mortality (participants affected / at risk) | 1/4 | 3/10 | 1/6 | 0/3 | 1/4 | 1/5 | 2/5 | 1/4 | 1/6 | 0/5 | 0/2 | 2/9 | 3/6 | 1/2 | 11/16 | 1/2 | 5/6 | 8/12
Serious Adverse Events (participants affected / at risk) | 3/4 | 7/10 | 3/6 | 2/3 | 4/4 | 2/5 | 4/5 | 2/4 | 2/6 | 3/5 | 1/2 | 2/9 | 4/6 | 2/2 | 9/16 | 2/2 | 3/6 | 6/12
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 6/6 | 3/3 | 4/4 | 5/5 | 5/5 | 4/4 | 6/6 | 5/5 | 2/2 | 8/9 | 5/6 | 2/2 | 15/16 | 2/2 | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: 50 mg Encorafenib QD (N=4) | Dose Escalation: 100 mg Encorafenib QD (N=10) | Dose Escalation:150 mg Encorafenib QD (N=6) | Dose Escalation: 75 mg Encorafenib BID (N=3) | Dose Escalation: 200 mg Encorafenib QD (N=4) | Dose Escalation: 100 mg Encorafenib BID (N=5) | Dose Escalation: 300 mg Encorafenib QD (N=5) | Dose Escalation: 150 mg Encorafenib BID (N=4) | Dose Escalation: 450 mg Encorafenib QD (N=6) | Dose Escalation: 550 mg Encorafenib QD (N=5) | Dose Escalation: 700 mg Encorafenib QD (N=2) | Dose Expansion: Mel Naive 300 mg Encorafenib (N=9) | Dose Expansion: Mel Naive 450 mg Encorafenib (N=6) | Dose Expansion: Mel Pre-treated 300 mg Encorafenib (N=2) | Dose Expansion: Mel Pre-treated 450 mg Encorafenib (N=16) | Dose Expansion: Mel Stepwise 450 mg Encorafenib (N=2) | Dose Expansion: Metastatic Colorectal Cancer 300 mg Encorafenib (N=6) | Dose Expansion: Metastatic Colorectal Cancer 450 mg Encorafenib (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: 50 mg Encorafenib QD (N=4) | Dose Escalation: 100 mg Encorafenib QD (N=10) | Dose Escalation:150 mg Encorafenib QD (N=6) | Dose Escalation: 75 mg Encorafenib BID (N=3) | Dose Escalation: 200 mg Encorafenib QD (N=4) | Dose Escalation: 100 mg Encorafenib BID (N=5) | Dose Escalation: 300 mg Encorafenib QD (N=5) | Dose Escalation: 150 mg Encorafenib BID (N=4) | Dose Escalation: 450 mg Encorafenib QD (N=6) | Dose Escalation: 550 mg Encorafenib QD (N=5) | Dose Escalation: 700 mg Encorafenib QD (N=2) | Dose Expansion: Mel Naive 300 mg Encorafenib (N=9) | Dose Expansion: Mel Naive 450 mg Encorafenib (N=6) | Dose Expansion: Mel Pre-treated 300 mg Encorafenib (N=2) | Dose Expansion: Mel Pre-treated 450 mg Encorafenib (N=16) | Dose Expansion: Mel Stepwise 450 mg Encorafenib (N=2) | Dose Expansion: Metastatic Colorectal Cancer 300 mg Encorafenib (N=6) | Dose Expansion: Metastatic Colorectal Cancer 450 mg Encorafenib (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 5 | 0 | 1 | 4 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 1 | 4 | 4 | 2 | 9 | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 3 | 2 | 3 | 2 | 2 | 7 | 2 | 5 | 2
Asthenia (General disorders) | 3 | 3 | 2 | 0 | 2 | 0 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 9 | 2 | 1 | 5
Chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 2 | 2 | 0 | 2 | 2 | 2 | 2 | 3 | 1 | 3 | 2 | 1 | 2 | 0 | 2 | 2
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Xerosis (General disorders) | 2 | 5 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 3
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 4 | 1 | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 0 | 3 | 2 | 0 | 1 | 4 | 1 | 4 | 1 | 2 | 3 | 0 | 1 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3 | 2 | 2 | 1 | 3 | 1 | 1 | 3 | 1 | 3 | 2 | 1 | 8 | 2 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 2 | 2 | 3 | 0 | 1 | 2 | 2 | 5 | 2 | 0 | 13 | 1 | 1 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 1 | 4 | 0 | 2 | 1 | 3 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 4 | 1 | 1 | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 0 | 2 | 2 | 0 | 2 | 2 | 2 | 1 | 4 | 0 | 0 | 9 | 1 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 10 | 1 | 1 | 5
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 1 | 2 | 2 | 1 | 1 | 2 | 2 | 0 | 5 | 2 | 0 | 8 | 0 | 1 | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 1 | 0 | 0 | 2 | 2 | 2 | 2 | 1 | 4 | 2 | 1 | 8 | 0 | 1 | 7
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 | 7 | 2 | 1 | 3 | 0 | 3 | 1 | 0 | 2 | 1 | 5 | 2 | 0 | 5 | 2 | 3 | 3
Hypotrichosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 3 | 2 | 0 | 3 | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 9 | 1 | 1 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 6 | 2 | 0 | 3 | 2 | 4 | 1 | 4 | 2 | 1 | 4 | 2 | 0 | 11 | 2 | 4 | 8
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 2
Papule (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7 | 2 | 1 | 1 | 3 | 2 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 6 | 2 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Oral hyperkeratosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.